CLINICAL TRIAL: NCT06621914
Title: The Effects of Different Blood Flow Restriction Training Methodologies During the Rehabilitation of Military Personnel With Lower Limb Musculoskeletal Injuries Primarily Limited by Pain: a 2 Part Randomised Controlled Trial (Phase One)
Brief Title: Is Low-load Resistance Training With Blood Flow Restriction Feasible During Rehabilitation of Military Personnel With Lower Limb Injuries? Phase One RCT.
Acronym: LIMITLESS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Defence Medical Rehabilitation Centre, UK (Other Government)
Collaborators: Northumbria University (Other)
Responsible Party: Principal Investigator, Peter Ladlow, Chief Investigator and Exercise Physiology Lead for UK Defence Rehabilitation, University of Bath
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2318/MODREC/24a
Record Dates: First submitted 2024-09-23; First posted 2024-10-01 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2024-11

CONDITIONS: Pain; Persistent Pain; Musculoskeletal Pain
Keywords: blood flow restriction; persistent pain; hypoalgesia
MeSH Terms: conditions — Pain; Musculoskeletal Pain | interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Intervention Model Description: The overall study is a two phase RCT. Phase one will investigate two different BFR-RT protocols (high- vs low-pressure) for 1-week (7x BFR-RT sessions in 5 days). Phase two will take the BFR-RT protocol that elicited the greatest improvement in symptoms (high- or low-pressure) and compare that to conventional Uk Defence Rehabilitation practices over a 3 week period (21x BFR-RT sessions over 15 days).
Masking Description: Due to the nature of the intervention, it is not possible to blind participants or outcome assessors to the treatment allocation. There is also no effective sham condition available. This is a common limitation within all blood flow restriction training research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BFR80 (Experimental): Low load blood flow restriction training with high-pressure cuff (80% AOP) in addition to standard residential rehabilitation consisting of; (1) exercise-based therapy delivered in group settings and individually to address a variety of physical components relating to their pathology (e.g., balance and co-ordination, cardiovascular endurance, mobility and flexibility, motor control and dynamic stability, and muscular strength), (2) patient education sessions (e.g., activity modification, behavioural change, and focusing on pain management), and (3) one-on-one support sessions (e.g., dietetics, occupational therapy, physiotherapy, podiatry, prosthesis/orthosis specialists, social workers, and speech and language therapists).
  Interventions: Device: BFR 80
- BFR40 (Active Comparator): Low load blood flow restriction training with low-pressure cuff (40% AOP) in addition to standard residential rehabilitation consisting of; (1) exercise-based therapy delivered in group settings and individually to address a variety of physical components relating to their pathology (e.g., balance and co-ordination, cardiovascular endurance, mobility and flexibility, motor control and dynamic stability, and muscular strength), (2) patient education sessions (e.g., activity modification, behavioural change, and focusing on pain management), and (3) one-on-one support sessions (e.g., dietetics, occupational therapy, physiotherapy, podiatry, prosthesis/orthosis specialists, social workers, and speech and language therapists).
  Interventions: Device: BFR40

INTERVENTIONS:
Device: BFR 80 — The intervention involves placing a pneumatic tourniquet system over the proximal thigh. The cuff is inflated to 80% of limb occlusion pressure during lower limb strengthening exercises. These exercises include leg press and knee extensor exercises. Four sets (30,15,15,15 repetitions) performed at 20% of one repetition maximum.
  Other Names: Blood flow restriction training; Occlusion training
  Arms: BFR80
Device: BFR40 — The intervention involves placing a pneumatic tourniquet system over the proximal thigh. The cuff is inflated to 40% of limb occlusion pressure during lower limb strengthening exercises. These exercises include leg press and knee extensor exercises. Four sets (30,15,15,15 repetitions) performed at 20% of one repetition maximum.
  Other Names: Blood flow restriction training; Occlusion training
  Arms: BFR40

SUMMARY:
Pain can be one of the primary limiting factors to progress following musculoskeletal injury and may be caused by trauma or degenerative changes. There are few exercise rehabilitation interventions able to relieve pain, thereby reducing the number of military personnel fit for operations. Low load blood flow restriction (BFR) exercise has been shown to elicit an analgesic response and promote beneficial physiological changes in a variety of clinical populations.

This two phase study, aims to:

* Determine the most effective and feasible BFR resistance exercise protocol for reducing pain in UK military patients.
* Determine the efficacy of an optimal BFR exercise protocol for reducing pain and improving rehabilitation outcomes in UK military patients.
* Identify key physiological mechanisms underpinning any beneficial effect of BFR exercise on pain.

Consequently, results from this study will have direct clinical application and will aid best practice guidelines for the management of pain across Defence Rehabilitation by influencing the future rehabilitation paradigm. The investigators believe the results and impact will be far reaching, providing invaluable insight and knowledge to the clinical and scientific community to not only those embedded within Defence Rehabilitation, but also those working in civilian sector organisations and professional sport also.

ELIGIBILITY:
Inclusion Criteria:

* Serving UK military personnel,
* Aged 18-55,
* Has unilateral lower limb injury whereby pain is the primary limiting factor hindering progression, as diagnosed by relevant consultant and team,
* Reduced occupational employability and function,
* Scheduled to attend DMRC Stanford Hall for 3 week residential rehabilitation course.

Exclusion Criteria:

MSK-Specific Exclusion Criteria

* Any medical contraindication related to BFR*
* Non-musculoskeletal or serious pathological condition (i.e. Inflammatory arthropathy, infection or tumour)
* Spinal or referred pain from non-local pain source
* Any pre-diagnosed physical impairment or co-morbidities (including cardio-vascular disease) precluding the safe participation in the rehabilitation programme and/or assessment procedures
* Corticosteroid or analgesic injection intervention to the affected area within the previous 7 days
* Currently pregnant, or have not yet completed a return to work assessment following the birth of your child.

  *Medical-Related Exclusion Criteria
* History of cardiovascular disease (hypertension, peripheral vascular disease, thrombosis/embolism, ischaemic heart disease, myocardial infarction),
* History of the following musculoskeletal disorders: rheumatoid arthritis, avascular necrosis or osteonecrosis, severe osteoarthritis
* History of the following neurological disorders: Alzheimer's disease, amyotrophic lateral sclerosis, peripheral neuropathy, Parkinson's disease, severe traumatic brain injury,
* Varicose veins in the lower limb,
* Acute viral or bacterial upper or lower respiratory infection at screening,
* Known or suspected lower limb chronic exertional compartment syndrome (CECS) (tourniquet raises intra-compartmental muscle pressure),
* Surgical insertion of metal components at the position of cuff inflation,
* History of any of the following conditions or disorders not previously listed: diabetes, active cancer,
* History of elevated risk of unexplained fainting or dizzy spells during physical activity and/or exercise that causes loss of balance,
* Increased risk of haemorrhagic stroke, exercise induced rhabdomyolysis,
* Currently pregnant.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-10-28 (Actual); Primary Completion 2026-05-29 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Brief Pain Inventory | Pre-intervention (day 0), post-intervention (day 5) and at follow-up (day 8).
  The BPI is a patient administered, multi-dimensional, pain assessment tool commonly used within musculoskeletal clinical practice. Higher scores on the 9-item short form indicate greater interference with function, or greater pain intensity.

SECONDARY OUTCOMES:
Pressure Pain Threshold Testing | Pre-intervention (day 0), daily (before, immediately-post, and 1hr-post each BFR session; days 1-5), post-intervention (day 5) and at follow-up (day 8).
  Pressure pain threshold assessment can help define regions of mechanical hypersensitivity, a common trait of central sensitisation. By utilising a digital pressure algometer (1cm^2 probe, Model FPX 50, Wagner Instruments, USA), the amount of pressure at which the sensation of pressure becomes unpleasant is deemed the PPT, with lower pressure values being indicative of central sensitisation.
Lower Extremity Function Scale | Pre-intervention (day 0), post-intervention (day 5) and at follow-up (day 8).
  The LEFS is a patient-reported outcome measure that measures functional status in patients with lower limb musculoskeletal injury. Ability to perform 20 activities, ranging from walking to running on uneven ground, are self-reported from 0-4 with higher scores indicating better function.
Isometric Mid-Thigh Pull | Pre-intervention (day 0), post-intervention (day 5) and at follow-up (day 8).
  The isometric mid-thigh pull is a test that can assess multiple derivatives of maximal lower-limb muscle strength including, peak force, rate of force development and limb asymmetry. The participant is asked to stand on force plates (set within a mid-thigh pull rig) and then pull on the mid-thigh bar at maximal force.
5-RM Testing | Pre-intervention (day 0) and follow-up (day 8).
  5-RM assessment on leg press and leg/knee extension machines (leg/knee extension pre-intervention only) to assess the participants strength, and inform % load for intervention period.
  Testing procedure: 5-minute cycling warm up, followed by 10-rep exercise specific warm up, and then successive attempts at performing a 5RM on injured limb only.
  The authors acknowledge that due to the likely interference effect of a pain response, performing a 'maximum effort' physical task in a lower limb injured cohort is unlikely to yield a true measure of MSK performance. It is more accurate to describe outcome scores as providing an 'indication' of participant performance and progression. We will highlight this as a potential weakness in our study but feel this is a challenge in the measurement of muscle force / strength in all MSK injury research. All outcomes measured will be implemented and recorded based upon a best effort at the time of assessment.
Numerical Pain Rating Scale | Daily (before, immediately-post, and 1 hour-post each BFR session; days 1-5).
  To assess the feasibility and tolerability of the BFR-RT interventions, a participant monitoring booklet will be used throughout the intervention period.
  The Numerical Pain Rating Scale (NPRS) for injury-specific pain and localised muscle soreness will be collected pre-intervention, immediately post-intervention, and 1-hour post-intervention for each BFR-RT session.
Sessional Rate of Perceived Exertion | Daily (immediately post-intervention; day 1-5).
  To assess the feasibility and tolerability of the BFR-RT interventions, a participant monitoring booklet will be used throughout the intervention period.
  Sessional Rate of Perceived Exertion (scored 0-10; 0=no effort, 10=maximal effort) will be collected following each BFR-RT session.
Training Load | Daily (immediately post-intervention; day 1-5).
  To assess the feasibility and tolerability of the BFR-RT interventions, a participant monitoring booklet will be used throughout the intervention period.
  To quantify training load, the following calculation will be conducted following each BFR-RT session; sets x reps x load (kg).
  Specific Example:
  BFR-RT Leg Press at 25kg
  1 set x 30 reps + 3 sets x 15 reps = 75 reps 75 (reps) x 25 (kg) = 1875 (training load)
Copenhagen Hip and Groin Score | Pre-intervention (day 0), post-intervention (day 5) and at follow-up (day 8).
  A single injury-specific outcome measure will also be collected at Day 0, Day 5 and Day 8.
  The Copenhagen Hip and Groin Score is a patient administered, multi-dimensional, pain assessment tool commonly used to assess symptomatic and functional burden associated with hip and groin pathology. Scored from 0-100, lower scores on the HAGOS represent greater symptomatic and functional burden. The MCID per domain is 8, 8, 9, 10, 11, and 12 points for hip-related QOL, symptoms, pain, sport and recreation activities, ADL, and participation in physical activities, respectively.
Foot and Ankle Disability Index | Pre-intervention (day 0), post-intervention (day 5) and at follow-up (day 8).
  A single injury-specific outcome measure will also be collected at Day 0, Day 5 and Day 8.
  The Foot and Ankle Disability Index is a 26-item ankle and foot specific, patient-reported, questionnaire which considers ADLs, function, pain and sleep. Each item is scored from 0 (unable to do/unbearable pain) to 4 (no difficulty at all/no pain), with a total point value reaching a maximum of 104; however, the PROM is scored as a percentage and a lower percentage indicates greater levels of disability and/or pain. To date, no MCID has been reported for the Foot and Ankle Disability outcome measure.
Leeds Assessment of Neuropathic Symptoms and Signs | Pre-intervention (day 0), post-intervention (day 5) and at follow-up (day 8).
  A single injury-specific outcome measure will also be collected at Day 0, Day 5 and Day 8.
  The Leeds Assessment of Neuropathic Symptoms and Signs is a self-reported questionnaire with a primary aim of distinguishing pain of a neuropathic origin, without the need for clinical assessment. The questionnaire consists of 7 questions, with a higher score suggesting the pain is predominantly of neuropathic origin. To date, no MCID has been reported for the Leeds Assessment of Neuropathic Symptoms and Signs.
Non-Arthritic Hips Score | Pre-intervention (day 0), post-intervention (day 5) and at follow-up (day 8).
  A single injury-specific outcome measure will also be collected at Day 0, Day 5 and Day 8.
  The Non-Arthritic Hips Score is a 20-item, self-reported, questionnaire covering four domains (activities, function, pain and symptoms), in patients without arthritic pathology. The summative score for Non-Arthritic Hips Score is between 0-100, with 100 representing a perfectly functioning hip. The MCID for this outcome measure is 8-points.
Victorian Institute for Sport Assessment - Gluteal | Pre-intervention (day 0), post-intervention (day 5) and at follow-up (day 8).
  A single injury-specific outcome measure will also be collected at Day 0, Day 5 and Day 8.
  The Victorian Institute for Sport Assessment - Glutealwas designed to evaluate the severity of disability in greater trochanteric pain syndrome populations. Formulated in the same manner as other Victorian Institute of Sport Assessment tendinopathy measures, the Victorian Institute for Sport Assessment - Gluteal is scored out of 100, with a greater score associated with greater function and less symptom impairment. There is currently no MCID reported within the literature for the Victorian Institute for Sport Assessment - Gluteal.
Victorian Institute for Sport Assessment - Hamstring | Pre-intervention (day 0), post-intervention (day 5) and at follow-up (day 8).
  A single injury-specific outcome measure will also be collected at Day 0, Day 5 and Day 8.
  The Victorian Institute for Sport Assessment - Hamstring was designed in the style of previous Victorian Institute of Sport Assessment tendinopathy outcome measures, but specifically to evaluate the severity of symptoms, function and ability to play sports in those with proximal hamstring tendinopathy. Scored out of 100, with higher scores being associated with greater function and less symptomatic impairments. A 4-point reduction was reported in the literature as being the threshold required to detect for true change when the standard error of measurement is considered; however, an MDIC of 22-points has been reported.
Victorian Institute for Sport Assessment - Patella | Pre-intervention (day 0), post-intervention (day 5) and at follow-up (day 8).
  A single injury-specific outcome measure will also be collected at Day 0, Day 5 and Day 8.
  The Victorian Institute for Sport Assessment - Patella is an 8 question, patient-reported measure developed specifically to subjectively assess the severity of symptoms, function and ability to play sports in those with patella tendinopathy . Scored out of 100, a greater score is associated with greater function and less symptom impairment, with 0 being the theoretical minimum score. The MCID for the Victorian Institute for Sport Assessment - Patella is 13-points.
Daily Morning Wellbeing | T2, Daily (before BFR session; days 1-5).
  To assess the feasibility and tolerability of the BFR-RT interventions, a participant monitoring booklet will be used throughout the intervention period.
  Daily morning wellbeing questions (fatigue, muscle soreness, sleep quality, stress levels and mood) will be asked each morning on a Likert scale (1-5), before the first BFR-RT session.
Knee Injury and Osteoarthritis Outcome Score | Pre-intervention (day 0), post-intervention (day 5) and at follow-up (day 8).
  A single injury-specific outcome measure will also be collected at Day 0, Day 5 and Day 8.
  The Knee Injury and Osteoarthritis Outcome Score is a five domain, patient-administered questionnaire, used to monitor disease course and outcomes following knee injury/OA or surgery. The five domains, ADL, knee-related QOL, other symptoms, pain, and sport and recreation function, are scored on a 0-100 scale, with a higher score indicating better function and less symptoms. The MCID for the Knee Injury and Osteoarthritis Outcome Score is 10-points for each domain.
Victorian Institute for Sport Assessment - Achilles | Pre-intervention (day 0), post-intervention (day 5) and at follow-up (day 8).
  A single injury-specific outcome measure will also be collected at Day 0, Day 5 and Day 8.
  The Victorian Institute for Sport Assessment - Achilles is a patient-reported questionnaire designed to assess the severity of Achilles tendinopathy. With questions focused on the domains of function in ADLs, pain, and sporting activity, the questionnaire is scored out of 100 (100 = asymptomatic); however, a score less than 60 is often seen in Achilles tendinopathy populations. The MCID is set at 14-points for mid-portion Achilles tendinopathy, and 6.5 points for insertional tendinopathy.
Musculoskeletal Health Questionnaire | T0, Pre-Admission (Day 0).
  The MSK-HQ is a self-reported questionnaire that allows people with musculoskeletal conditions to report their symptoms and quality of life in a standardised way. This outcome measure is taken at baseline only (T0).
Health Anxiety Depression Scale | T0, Pre-Admission (Day 0).
  The Hospital Anxiety and Depression Scale (HADS) is a 14-item self-reported measure designed to assess anxiety and depression symptoms in medical patients, with emphasis on reducing the impact of physical illness on the total score. This outcome measure is taken at baseline only (T0).
Demographics Questionnaire | T0, Pre-Admission (Day 0).
  Personal and demographic characteristics including age, body height, body mass, body mass index, duration of symptoms, previous injuries, previous treatment, military occupation, duration of military service, smoking and drinking habits. This outcome measure is taken at baseline only (T0).
Medication Record Sheet | T0, Pre-Admission (Day 0).
  The medication record sheet is utilised to show what current medications each participant is using for their pathology. The drug name, drug purpose, dose size and frequency is noted. This outcome measure is taken at baseline only (T0).

CONTACTS AND LOCATIONS:
Overall Officials: Peter Ladlow, PhD, Principal Investigator — Defence Medical Rehabilitation Centre, UK
Locations (1):
- Defence Medical Rehabilitation Centre, Stanford Hall, Loughborough, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Upon reasonable request, grouped data (i.e., data that cannot individually identify participants) may be shared to other research groups for the advancement of research and clinical practices, by the chief investigator.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Upon completion of the dissemination of research findings (i.e., publications and conference proceedings).
Access Criteria: Most data will be openly available, but due to privacy concerns, some data regarding participants are available only to bona fide researchers working on a related project, subject to the completion of a non-disclosure agreement.

REFERENCES:
- [Derived] Gray L, Coppack RJ, Barker-Davies R, Cassidy RP, Bennett AN, Caplan N, Atkinson G, Bradshaw L, Chauhan J, Lunt KM, Hughes L, Ladlow P. Efficacy and acceptability of different blood flow restriction training interventions during the rehabilitation of military personnel with lower limb musculoskeletal injuries: protocol for a two-phase randomised controlled trial. BMJ Open. 2025 May 26;15(5):e096643. doi: 10.1136/bmjopen-2024-096643. PMID 40425246